CLINICAL TRIAL: NCT04684914
Title: Phase 2, Double-blind, Randomized, Placebo-controlled Study of HepTcell (Adjuvanted FP-02.2) as an Immunotherapeutic Vaccine in Treatment-naïve Patients With Inactive Chronic Hepatitis B (CHB)
Brief Title: HepTcell Immunotherapy in Patients With Inactive Chronic Hepatitis B (CHB)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Did not meet endpoints
Sponsor: Altimmune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALT-301-202
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Results first posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Hepatitis B, Chronic
Keywords: Immunotherapy; CHB
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HepTcell (Experimental): Dose administered at intervals of 4 weeks for 6 doses
  Interventions: Biological: HepTcell
- Placebo (Placebo Comparator): Dose administered at intervals of 4 weeks for 6 doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: HepTcell — Intramuscular injection
  Arms: HepTcell
Drug: Placebo — Intramuscular injection
  Arms: Placebo

SUMMARY:
A study to evaluate the antiviral effects, immunogenicity, and safety of HepTcell in treatment-naive patients with inactive chronic hepatitis B (CHB) and low hepatitis B surface antigen (HBsAg) levels.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 to 65 years of age, inclusive
* Inactive CHB with documented HBsAg positivity for at least 12 months before Day 1
* qHBsAg ≥ 10 IU/mL but ≤ 100 IU/mL in the 12 months prior to screening
* HBV DNA ≥ 10 IU/mL at screening
* AST, ALT, INR, albumin, total bilirubin (excluding patients with Gilbert Syndrome) and direct bilirubin within normal limits at screening

Exclusion Criteria:

* Positive hepatitis B e antigen (HBeAg) at screening
* History of a hepatitis B flare or 1-log increase in HBV DNA or HBsAg in the prior 12 months
* Undetectable HBV DNA at screening
* Fibroscan > 8.5 kPA at screening, or history of hepatic fibrosis or cirrhosis (NB, a Fibroscan is not required if an examination is performed within 12 months or a liver biopsy was performed within 2 years before Screening and no fibrosis [F1 or greater] was identified).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2020-12-26 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-04-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (5):
  - Paragon Rx Clinical, Garden Grove, California
  - Stanford University Department of Medicine, Redwood City, California
  - San Jose Gastroenterology Institute, San Jose, California
  - Kansas City Research Institute, Kansas City, Missouri
  - Central Sooner Research, Oklahoma City, Oklahoma
- Canada (5):
  - University of Calgary Liver Unit - Heritage Medical Research Clinic, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - The Ottawa Hospital, Ottawa, Ontario
  - Toronto Centre for Liver Disease (TCLD), Toronto General Hospital, UHN, Toronto, Ontario
  - Toronto Liver Centre, Toronto, Ontario
- Germany (2):
  - Goethe University Hospital, Frankfurt am Main
  - Univesritätsklinikum Hamburg-Eppendorf, Hamburg
- Spain (6):
  - Hospital Clínic De Barcelona, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Nuestra Señora De Valme, Seville
  - Consorcio Hospital General Universitario De Valencia, Valencia
  - Hospital Universitari I Politècnic La Fe, Valencia
- United Kingdom (3):
  - St. Georges University of London, London
  - St. Mary's Hospital, London
  - Queens Medical Center, Nottingham

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HepTcell | Placebo
Started | 42 | 45
Treated (One subject randomized to HepTcell and 2 subjects randomized to placebo discontinued before receiving study treatment) | 41 | 43
Completed | 40 | 43
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Discontinued before receiving study treatment | 1 | 2

BASELINE CHARACTERISTICS:
Population: mITT population: all randomized subjects who received any amount of study medication and had a baseline and at least one postbaseline efficacy assessment
Groups:
- Total: Total of all reporting groups
Arm/Group | HepTcell | Placebo | Total
Number analyzed (Participants) | 41 | 43 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.95 (9.07) | 53.21 (8.08) | 52.11 (8.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 19 | 32
  Male | 28 | 24 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 27 | 24 | 51
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 6 | 8
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 6 | 8 | 14
  United States | 6 | 4 | 10
  United Kingdom | 1 | 4 | 5
  Germany | 0 | 1 | 1
  Spain | 9 | 11 | 20
  Thailand | 13 | 12 | 25
  Italy | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients Achieving Virologic Responses
Description: Virologic response is defined as a 1.0-log reduction in quantitative hepatitis B surface antigen (HBsAg) or serologic clearance of HBsAg from Baseline to Day 169
Time Frame: Baseline to Day 169
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | HepTcell | Placebo
Number analyzed (Participants) | 41 | 43
Participants | 1 | 0
Statistical Analysis 1: Comparison: HepTcell vs Placebo; Test type: Superiority; p = 0.3029, Chi-squared
Statistical Analysis 2: Comparison: HepTcell vs Placebo; Test type: Superiority; p = 0.4881, Fisher Exact

2. Secondary Outcome: The Proportion of Patients Achieving Serologic Clearance of Hepatitis B Surface Antigen (HBsAg) on Day 169
Time Frame: Baseline to Day 169
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | HepTcell | Placebo
Number analyzed (Participants) | 41 | 43
Participants | 1 | 0
Statistical Analysis 1: Comparison: HepTcell vs Placebo; Test type: Superiority; p = 0.3029, Chi-squared
Statistical Analysis 2: Comparison: HepTcell vs Placebo; Test type: Superiority; p = 0.4881, Fisher Exact

3. Secondary Outcome: The Proportion of Patients Achieving Serologic Clearance of Hepatitis B Virus (HBV) DNA on Day 169
Time Frame: Baseline to Day 169
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | HepTcell | Placebo
Number analyzed (Participants) | 41 | 43
Participants | 5 | 8
Statistical Analysis 1: Comparison: HepTcell vs Placebo; Test type: Superiority; p = 0.4169, Chi-squared
Statistical Analysis 2: Comparison: HepTcell vs Placebo; Test type: Superiority; p = 0.5495, Fisher Exact

4. Secondary Outcome: Changes in Quantitative HBsAg Level
Time Frame: Baseline to Days 85 and 169
Population: mITT. Number analyzed are the number of participants with data at each time point. Changes from baseline are calculated only for participants with non-missing values for both the baseline and time point of interest.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | HepTcell | Placebo
Number analyzed (Participants) | 41 | 43
IU/mL
  Day 85: number analyzed (Participants) | 40 | 43
  Day 85 | -7.76 (28.01) | -8.47 (15.85)
  Day 169 | -13.72 (32.80) | -10.19 (31.87)

5. Secondary Outcome: Changes in HBV DNA Levels
Time Frame: Baseline to Days 85 and 169
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | HepTcell | Placebo
Number analyzed (Participants) | 41 | 43
IU/mL
  Day 85: number analyzed (Participants) | 37 | 39
  Day 85 | -7559.73 (46650.54) | -5270.05 (33240.79)
  Day 169: number analyzed (Participants) | 40 | 42
  Day 169 | -7868.48 (44871.40) | -4690.12 (32070.75)

6. Secondary Outcome: Changes in Hepatitis B Core-related Antigen (HBCrAg) Levels
Time Frame: Baseline to Days 85 and 169
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kU/mL
Arm/Group | HepTcell | Placebo
Number analyzed (Participants) | 41 | 43
kU/mL
  Day 85: number analyzed (Participants) | 3 | 1
  Day 85 | -4.00 (7.81) | 1.00 (NA) — Data from a single subject
  Day 169: number analyzed (Participants) | 3 | 1
  Day 169 | -1.00 (1.00) | 1.00 (NA) — Data from a single subject

7. Secondary Outcome: Changes in Pre-genomic RNA Levels
Time Frame: Baseline to Days 85 and 169
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Log U/mL
Arm/Group | HepTcell | Placebo
Number analyzed (Participants) | 41 | 43
Log U/mL
  Day 85: number analyzed (Participants) | 17 | 17
  Day 85 | 0.26 (0.42) | 0.16 (0.39)
  Day 169: number analyzed (Participants) | 17 | 17
  Day 169 | 0.31 (0.44) | 0.30 (0.48)

8. Secondary Outcome: Change in IFN-gamma Frequency by ELISpot Assay in PBMCs
Description: Percent change in antigen-specific spot forming cells per million peripheral blood mononuclear cells (PBMCs)
Time Frame: Baseline to Days 85 and 169
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | HepTcell | Placebo
Number analyzed (Participants) | 41 | 43
percent change
  Day 85: number analyzed (Participants) | 40 | 43
  Day 85 | 3.71 (39.02) | -0.14 (21.50)
  Day 169 | -5.28 (28.56) | 3.45 (45.56)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | HepTcell | Placebo
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/43
Other Adverse Events (participants affected / at risk) | 19/41 | 29/43
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HepTcell (N=41) | Placebo (N=43)
COVID-19 (Infections and infestations) | 6 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Headache (Nervous system disorders) | 2 | 2
Pyrexia (General disorders) | 2 | 2
Neutrophil count decreased (Investigations) | 1 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 2
Food poisoning (Gastrointestinal disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Influenza A virus test positive (Investigations) | 0 | 2
Fatigue (General disorders) | 0 | 2
Limb injury (Injury, poisoning and procedural complications) | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Iron deficiency (Metabolism and nutrition disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-07-24): https://cdn.clinicaltrials.gov/large-docs/14/NCT04684914/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT04684914/SAP_001.pdf